# Computed Tomography Coronary Angiography (CTCA) prior to Chronic Total Occlusion (CTO) Percutaneous Coronary Intervention (PCI) - a feasibility study

## **TRIAL SUMMARY**

| Trial Title | Computed Tomography Coronary Angiography (CTCA) |
|---|---|
| | prior to Chronic Total Occlusion (CTO) Percutaneous |
| | Coronary Intervention (PCI) - a feasibility study |
| Summary of Trial design | Randomised, prospective, single centre feasibility study of |
| | CTCA prior to CTO PCI |
| Site and Chief Investigator | Sandwell and West Birmingham NHS Trust, Birmingham, |
| | United Kingdom |
| | Vinoda Sharma |
| Participant population | Patients undergoing CTO PCI |
| Planned sample size | 20 |
| Number of sites | 1 |
| Intervention duration | Prior to index CTO PCI procedure |
| Follow up duration | 6 months |
| Planned trial duration | 1 year |
| Primary objective | To determine if CTCA prior to CTO PCI results in improved procedural success rate? |
| Secondary objectives | i) To determine if CTCA prior to CTO PCI results in improved angina as determined by Seattle Angina Questionnaire (SAQ)? ii) To determine if CTCA prior to CTO PCI reduces the need for a second procedure due to improved procedural success rate? iii) Are there procedural differences between the intervention arm (CTCA) and usual care |
| Intervention | Randomised to CTCA versus no CTCA prior to CTO PCI |

### **ABBREVIATIONS:**

**CABG:** Coronary Artery Bypass Graft

**CAD:** Coronary Artery Disease

**CTCA:** Computed Tomography Coronary Angiogram

CTO: Chronic Total Occlusion

**J-CTO:** Japanese Chronic Total Occlusion

**PCI:** Percutaneous Coronary Intervention

**QALYS:** Quality Adjusted Life Years

QoL: Quality of Life

**SAQ:** Seattle Angina Questionnaire

## **Trial Protocol Synopsis**

| Computed Tomography Coronary Angiography (CTCA) prior to Chronic Total Occlusion (CTO) Percutaneous Coronary Intervention (PCI) |
|---|
| to Chronic Total Occlusion (CTO) Percutaneous Coronary |
| Null Hypothesis: CTCA performed prior to CTO PCI will not improve procedural success |
| Existing knowledge: A chronic total occlusion (CTO) is present in 15-20% of patients with angina who are referred for coronary angiography. Due to the complexity of occlusive coronary artery disease (CAD), including a high prevalence of calcium and tortuosity within long segments of disease, CTO PCI is associated with higher procedural complication rates (11). Inability to detect the intraluminal path in the CTO artery, combined with calcification and tortuosity can result in unsuccessful guidewire crossing and procedural failure. Successful CTO PCI has been shown to improve Quality of Life (QoL) at 12 months(4). These patients are more likely to be angina free at 12 months (5, 6) as assessed by the Seattle Angina Questionnaire (SAQ) (7, 8). CTO PCI in symptomatic patients is cost effective and results in greater quality-adjusted-life-years (QALYS)(9, 10). |
| CTO percutaneous coronary intervention (PCI) procedure success rates increased from 68% to 79% between 2000 and 2011, and are as high as 90% when performed by high-volume CTO operators (2, 3). Complexity of the CTO is determined by several factors and several CTO complexity scores, derived from (invasive) angiographic lesion and clinical characteristics, have been shown to correlate with procedural success and complication rates (JCTO(12), PROGRESS(13), RECHARGE(14), Euro-CASTLE(15)). The most commonly utilised score is the J-CTO (Multicenter Chronic Total Occlusion Registry of Japan)(12) which assigns a score of 1 each to the angiographic CTO proximal cap (tapered or blunt), calcification, tortuosity (>45°), lesion length (≥20mm) and previous failure, with a maximum score =5. Scores ≥2 are considered CTOs that are difficult to perform and require advanced techniques for successful revascularisation. In a proportion of these patients, the first procedure either fails completely or partially succeeds in forming a tract within the occluded artery but this is inadequate for stent delivery and the patient requires a second procedure, |

reconstruction of the fully occluded artery.

Angiographically, the CTO artery usually shows a short proximal portion of dye filled artery prior to the occlusion. In most patients there are some collaterals from the contralateral coronary artery which try to fill part of the occluded CTO artery. However the actual body of the CTO is not visible angiographically.

Computed Tomography Coronary Angiography (CTCA) can delineate the coronary anatomy in 3-dimensions, determining atherosclerotic plaque and occlusion location, severity and morphology. This makes it an attractive modality to assess the coronary CTO. Development of a CTCA based complexity score for stratifying CTOs by difficulty resulted in the CT-RECTOR score (Computed Tomography Registry of Chronic Total Occlusion Revascularization, table 1)(16). Variables included in this score are multiple occlusions, blunt stump, severe calcification, bending, duration of CTO ≥12 months and previously failed PCI (all scored 1). The CT-RECTOR score correlates with the J-CTO score and has a better area under ROC curve (ROC AUC 0.83 for CT-RECTOR score and 0.71 for J-CTO, p < 0.001) and predicts CTO PCI success (16)

The role of routine CTCA pre-CTO PCI is as yet undefined as current practice involves the use of CTCA in patients who have had an unsuccessful CTO PCI attempt or previous coronary artery bypass grafting (CABG).

#### Need for a feasibility study:

Current practice at our centre involves the use of CTCA in patients who have had an unsuccessful CTO PCI attempt or previous coronary artery bypass grafting (CABG) but the role of routine CTCA pre-CTO PCI is as yet undefined.

The small additional investment of a CTCA could help plan/improve a complex procedure and may reduce the need for additional procedures and readmissions.

The mean acute treatment cost of a CTO PCI is approximately (combined day-case –ordinary elective spell) £6933 (9, 17) whereas the approximate cost of a CTCA is £360 (as per local billing). Elective readmission for a failed CTO PCI procedure would entail an additional financial (to the provider) and emotional cost (to the patient).

The cost of an additional CTO PCI procedure aside, readmission and bed charges themselves can reach £1000/day (readmission =£255/day)(17)and bed

| | cost=£600/day). Including the cost of a second CTO PCI procedure (combined day-case –ordinary elective spell) £6933 (9, 17), the overall cost can total to £10,000. In contrast, the cost of a CTCA is £360 (as per local billing). Financial costs are one part of the issue, but a second CTO PCI procedure can also heighten patient anxiety and discomfort which are well known in patients prior to any PCI. |
|---|---|
| | A feasibility study will help establish the role of a CTCA prior to CTO PCI to positively influence strategy and/or outcomes. |
| Objectives | Primary: |
| | i) Does performing a CTCA prior to CTO PCI<br>improve the success of the CTO procedure? |
| | Secondary: |
| | i) To determine if CTCA prior to CTO PCI results in improved angina as determined using the Seattle Angina Questionnaire (SAQ) by SAQ. |
| | ii) To determine if CTCA prior to CTO PCI reduces the need for a second procedure (due to improved procedural success rate). |
| | iii) To assess if there are procedural differences between the intervention arm (CTCA) and usual care arm |
| Comparators | CTCA versus no CTCA prior to CTO PCI |
| Trial design | Randomised (1:1), prospective, single centre study |
| Methods (see figure 1) | |
| Study setting | Sandwell and West Birmingham NHS Trust, Birmingham, United Kingdom |
| Eligibility Criteria | <ul> <li>Inclusion Criteria:</li> <li>Patients meeting all the below criteria will be included</li> <li>≥18 years</li> <li>CTO with J-CTO score≥2</li> <li>Appropriate indication for CTO PCI</li> <li>Adequate CTCA images for analysis</li> </ul> |
| | Exclusion criteria: Patients meeting any of the following criteria will be excluded • <18 years of age |
| | <ul><li>CTO with J-CTO score&lt;2</li><li>Inadequate/degraded CTCA images</li></ul> |
| | <ul> <li>Pregnant/lactating women</li> <li>Patients with severe contrast allergy</li> </ul> |
| | <ul> <li>Patients unable to provide written informed<br/>consent</li> </ul> |

| Intervention | Experimental group: CTCA prior to CTO PCI Conventional group: CTO PCI Patients will be randomised to CTCA or no CTCA prior to |
|---|---|
| Outcomes | CTO PCI (figure 1) |
| Participant/project timeline | Outcomes Primary endpoint i. CTO PCI success rate in CTCA arm versus no CTCA arm Secondary endpoints i. Angina by the SAQ summary score at 6 months ii. Compare the number of patients who required a second CTO PCI procedure in the CTCA arm versus no CTCA arm iii. Procedural differences between the intervention CTCA arm versus no CTCA arm including: a) Health Economics: • Cost saved per patient due to improved success and reduction in readmission or further procedure b) CTO PCI efficiency: • Wire crossing time • Procedure time c) CTO PCI safety outcomes: • Procedural complications (Ellis perforation, tamponade, acute kidney injury/contrast induced nephropathy, access site bleeding, donor vessel injury) • Radiation: CTCA dose, CTO PCI dose, and combined CTCA and CTO PCI dose, and combined CTCA and CTO PCI volume, and combined CTCA and CTO PCI volume, and combined CTCA and CTO PCI volume d) Change in CTO PCI strategy hierarchy as a result of the CTCA review |
| Sample size | This is a feasibility study- to ensure completion within a year, we have estimated 20 patients, randomised 1:1 to |
| | each arm (10 patients per arm) as a sample size in a moderate size hospital which performs approximately 100 CTO PCIs annually |
| Intervention assignment | Block randomisation with sealed envelope technique |
| Data collection, management and analysis | <ul> <li>eCRF and online database to collect demographic,<br/>procedural and SAQ information</li> </ul> |

| | <ul> <li>SAQ summary score at 6 months post PCI</li> <li>Blood samples pre and post PCI</li> <li>Comparison of demographics, procedural details, procedural success and complications, bloods, SAQ, and financial cost between the CTCA and non-CTCA groups</li> <li>Categorical variables will be presented as percentage and compared with the chi square or Fisher's test</li> <li>Continuous variables will be presented as median (range) and compared with student's t-test or Mann Whitney test.</li> <li>In addition, modelling will be performed by binary logistic regression analysis to predictors of CTO PCI success.</li> </ul> |
|---|---|
| Monitoring | CTO PCI procedural adverse events will be reported as usual on the national database and this data will be collected in the eCRF. |
| Ethics | Ethical approval for this prospective study will be obtained All patients will be consented prior to inclusion in this study |
| Blood | Routine blood tests will be performed immediately before the CTO PCI and after the procedure prior to discharge as standard of care |

Symptomatic CTO patients n=20 SAQ initial in all patients Ī Routine blood tests 1:1 randomisation to CTCA pre and post procedure No CTCA CTCA prior to CTO PCI SAQ final 6 months post-procedure CTO PCI CTO PCI in all patients

Figure 1: Patient flow pathway

Figure 2: Participant/project Timeline



#### **References:**

- 1. Opolski MP, Achenbach S. CT Angiography for Revascularization of CTO: Crossing the Borders of Diagnosis and Treatment. JACC Cardiovasc Imaging. 2015;8(7):846-58.
- 2. Patel VG, Brayton KM, Tamayo A, Mogabgab O, Michael TT, Lo N, et al. Angiographic success and procedural complications in patients undergoing percutaneous coronary chronic total occlusion interventions: a weighted meta-analysis of 18,061 patients from 65 studies. JACCCardiovascular interventions. 2013;6(2):128-36.
- 3. Sharma V, Jadhav ST, Harcombe AA, Kelly PA, Mozid A, Bagnall A, et al. Impact of proctoring on success rates for percutaneous revascularisation of coronary chronic total occlusions. Open Heart. 2015;2(1):e000228.
- 4. Simon W. The Consistent CTO Study. 2018.
- 5. Olivari Z, Rubartelli P, Piscione F, Ettori F, Fontanelli A, Salemme L, et al. Immediate results and one-year clinical outcome after percutaneous coronary interventions in chronic total occlusions: data from a multicenter, prospective, observational study (TOAST-GISE). J Am Coll Cardiol. 2003;41(10):1672-8.
- 6. Werner GS, Martin-Yuste V, Hildick-Smith D, Boudou N, Sianos G, Gelev V, et al. A randomized multicentre trial to compare revascularization with optimal medical therapy for the treatment of chronic total coronary occlusions. Eur Heart J. 2018;39(26):2484-93.
- 7. Chan PS, Jones PG, Arnold SA, Spertus JA. Development and validation of a short version of the Seattle angina questionnaire. Circ Cardiovasc Qual Outcomes. 2014;7(5):640-7.
- 8. Spertus JA, Winder JA, Dewhurst TA, Deyo RA, Prodzinski J, McDonell M, et al. Development and evaluation of the Seattle Angina Questionnaire: a new functional status measure for coronary artery disease. J Am Coll Cardiol. 1995;25(2):333-41.
- 9. Gada H, Whitlow PL, Marwick TH. Establishing the cost-effectiveness of percutaneous coronary intervention for chronic total occlusion in stable angina: a decision-analytic model. Heart. 2012;98(24):1790-7.
- 10. Grantham JA, Jones PG, Cannon L, Spertus JA. Quantifying the early health status benefits of successful chronic total occlusion recanalization: Results from the FlowCardia's Approach to Chronic Total Occlusion Recanalization (FACTOR) Trial. Circ Cardiovasc Qual Outcomes. 2010;3(3):284-90.
- 11. Tajti P, Brilakis ES. Chronic Total Occlusion Percutaneous Coronary Intervention: Evidence and Controversies. J Am Heart Assoc. 2018;7(2).
- 12. Morino Y, Abe M, Morimoto T, Kimura T, Hayashi Y, Muramatsu T, et al. Predicting successful guidewire crossing through chronic total occlusion of native coronary lesions within 30 minutes: the J-CTO (Multicenter CTO Registry in Japan) score as a difficulty grading and time assessment tool. JACCCardiovascular interventions. 2011;4(2):213-21.
- 13. Christopoulos G, Kandzari DE, Yeh RW, Jaffer FA, Karmpaliotis D, Wyman MR, et al. Development and Validation of a Novel Scoring System for Predicting Technical Success of Chronic Total Occlusion Percutaneous Coronary Interventions: The PROGRESS CTO (Prospective Global Registry for the Study of Chronic Total Occlusion Intervention) Score. JACC Cardiovasc Interv. 2016;9(1):1-9.
- 14. Maeremans J, Spratt JC, Knaapen P, Walsh S, Agostoni P, Wilson W, et al. Towards a contemporary, comprehensive scoring system for determining technical outcomes of hybrid percutaneous chronic total occlusion treatment: The RECHARGE score. Catheter Cardiovasc Interv. 2018;91(2):192-202.
- 15. Szijgyarto Z, Rampat R, Werner GS, Ho C, Reifart N, Lefevre T, et al. Derivation and Validation of a Chronic Total Coronary Occlusion Intervention Procedural Success Score From the 20,000-Patient EuroCTO Registry: The EuroCTO (CASTLE) Score. JACC Cardiovasc Interv. 2019;12(4):335-42.

- 16. Opolski MP, Achenbach S, Schuhbäck A, Rolf A, Möllmann H, Nef H, et al. Coronary computed tomographic prediction rule for time-efficient guidewire crossing through chronic total occlusion: insights from the CT-RECTOR multicenter registry (Computed Tomography Registry of Chronic Total Occlusion Revascularization). JACC Cardiovasc Interv. 2015;8(2):257-67.
- 17. Improvement N. 2019/20 National Tariff Payment System. 2019.

## Appendix

# Costing (approximate):

| Grade of staff/Test required | Role | Cost per patient | Work Time<br>Equivalent | Period of time | Total Cost all patients |
|---|---|---|---|---|---|
| CTCA per patient | - | £360/- | - | - | £7200 |
| Blood tests per patient | - | £30 per set x2<br>lots=£60 | | - | £1200 |
| Clinical<br>fellow/registrar | Patient consent,<br>review of blood<br>tests, telephone<br>follow up | - | | | £16,300 |
| Total | | | | | £24,700 |